CLINICAL TRIAL: NCT05457517
Title: A Multi-Center, Open-Label, Phase Ib/2 Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activity of YL-13027 Combined With Sintilimab in Patients With Advanced Solid Tumors
Brief Title: A Phase 1b/2 Study of YL-13027 Combined With Sintilimab in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai YingLi Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YL-13027-002
Record Dates: First submitted 2022-06-27; First posted 2022-07-14 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: YL-13027 combined with Sintilimab was used as a cycle for 21 days.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YL-13027+Sintilimab (Experimental): YL-13027 tablets will be given daily for 21 days in 21-day cycles until there appears evidence of progressive disease, intolerable toxicity, or the patient discontinues from the study treatment for other reasons.
  Sindilizumab injection will be given 200mg every three weeks.
  Interventions: Drug: YL-13027，Sintilimab

INTERVENTIONS:
Drug: YL-13027，Sintilimab — YL-13027 combined with Sintilimab will be used as a cycle for 21 days. YLl-13027 is administered orally twice a day. Starting dose of YL-13027 is 240mg/d，with escalation to 360mg/d in phase Ib, and RP2D was administered orally twice a day in phase II.
  Sindilizumab is administered intravenously 200mg every three weeks
  Other Names: YL-13027 tablet，Sintilimab injection

SUMMARY:
This study is a one-arm, open, multicenter phase 1b/2 clinical trial of YL-13027 combined with Sintilimab in patients with Advanced Solid Tumors, aiming at exploring the MTD and RP2D and observing the preliminary efficacy.The trial can be divided into two parts: dose escalation part and expansion part.Sintilimab is administered as a fixed-dose intravenous injection(200mgQ3w）.

DETAILED DESCRIPTION:
Part 1 (Phase Ib):

This is a dose escalation,3+3 design study, to evaluate the safety and tolerability, and to determine the RP2D of YL-13027 when administered b.i.d. in patients with advanced solid tumors. One cycle is 21 days.

Part 2 (Phase II):

This is an expansion phase in patients with advantage advanced solid tumors to further evaluate the safety, tolerability and preliminary anti-tumor activity of YL-13027 at the RP2D combined with Sintilimab.

ELIGIBILITY:
Inclusion Criteria:

1. Males and/or females age from 18 to 75.
2. Histologically or cytologically confirmed patients with advanced malignant solid tumors, extracranial solid tumors must be malignant tumors, including but not limited to lung cancer, head and neck cancer, renal clear cell carcinoma, urinary epithelial carcinoma, chordoma, etc. Intracranial primary tumors include malignant tumors and some benign tumors lacking effective standard treatment after current recurrence, including but not limited to glioma, meningioma, ependymoma, craniopharyngioma, refractory pituitary tumor, etc. Eligible patients must have failed standard treatment, have no standard treatment, have refused standard treatment, or have been determined by the investigator to be unsuitable for standard treatment at this stage.
3. At least 1 measurable lesion according to tumor assessment criteria.
4. Eastern Cooperative Oncology Group performance status of 0 to 2.
5. Life expectancy of at least 3 months.
6. Acceptable organ function: Absolute neutrophil count(ANC)≥1.5×109/L, Platelet count(PLT)≥100×109/L, Hemoglobin(Hb)≥90 g/L, Total bilirubin(TBIL)≤1.5×Upper limit of normal value(ULN), Alanine aminotransferase(ALT)≤2.5×ULN, Aspartate aminotransferase(AST)≤2.5×ULN, Creatinine(Cr)≤1.5×ULN, Creatinine clearance ≥50ml/min, Left Ventricular Ejection Fractions(LVEF)≥50%, QTcF<450 ms.
7. The washout period from the last time accepting any anti-tumor treatment (including chemotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy, tumor embolization) to participating in this test should be 3 weeks or more.The washout period of oral fluorouracil should be 2 weeks or more, and that of mitomycin and nitrosocarbamide should be 6 weeks or more.The washout period of drugs with anti-tumor angiogenic effects (those targeting VEGF, VEGF receptors including, but not limited to bevacizumab, anlotinib, apatinib, furquinib, lenvatinib, sorafenib, regorafenib, etc.) should be 8 weeks or more. The washout period of other anti-tumor treatments (radiotherapy, treatment with other test drugs) should be 4 weeks or more.
8. Fertile male and female must agree to use medically approved contraceptives during the study and within 6 months after the last dose of the study.
9. Blood pregnancy test of female who is capable of conceivingshould be negative 7 days before the first dose.Patients cannot breastfeed.If the patient has stopped breastfeeding at the time of study entry, the cessation of breastfeeding must be from the day of first dose to more than 30 days after the last dose.
10. The last time participate in an investigational drug study should be more than one month prior to the study entry.
11. According to the judgment of the investigator, the patient has high compliance and is willing to complete the experiment and comply with the protocol.
12. Voluntary participation in this clinical trial, understanding of the study procedures and the ability to sign informed consent forms (ICFs).

Exclusion Criteria:

1. There is third interstitial effusion (such as massive pleural effusion and ascites) which can not be controlled by drainage or other methods.
2. Within 3 months before the first dose, grade 3 or grade 4 gastrointestinal bleeding or varicose bleeding and requiring blood transfusion or endoscopic or surgical intervention has happened.
3. Medical history of difficulty in swallowing, malabsorption, or other chronic gastrointestinal disease, or conditions that may hamper compliance and/or absorption of the tested product.
4. Patients with a definitely history of neurological or psychiatric disorders.
5. Known infection with human immunodeficiency virus (HIV), hepatitis B virus(HBV), or hepatitis C virus (HCV).
6. History of immunodeficiency, including HIV positive test, other acquired or congenital immunodeficiency disorders, organ transplantation or allogeneic bone marrow transplantation.
7. Exists moderate or severe heart disease: (1) Within 6 months before the first dose,myocardial infarction, angina, grade II/III/IV congestive heart failure, pericardial effusion, uncontrollable severe hypertension (up to 150/90 mmHg or more) . (2) ECG abnormalities with clinical significance: symptomatic or persistent atrial or ventricular arrhythmias, degree II or III atrioventricular block, bundle branch block. (3) The echocardiogram shows significant abnormalities: For example, moderate or severe heart valve function defects are assessed according to the normal lower limit of the institution;Patients with minor or mild valve regurgitation (tricuspid, pulmonary, mitral, or aortic) can be included in this study. (4) Laboratory examination shows troponin T levels increasing. (5) Various factors that may increase the risk of QTcF prolonging or arrhythmia events. (6) Predisposition factors cause the development of ascending aorta or aortic arch aneurysm: For example, marfan syndrome, CT records of the history of cardiac vascular injury. (7) History of heart or aortic surgery.
8. Intracerebral lesions with significant space occupying effects (needing Dehydration treatment, glucocorticoid treatment or diuretic treatment)，spinal cord or pia mater dissemination.
9. At the beginning of the study, the unrecovered toxicity of the previous treatment exceeded CTCAE5.0 grade 1(except for hair loss).
10. According to the judgement of the researcher,there are concomitant diseases that seriously endanger the safety of patients or affect the completion of the study (such as severe hypertension, diabetes, thyroid diseases, etc.).
11. Patients has received vaccines other than inactivated vaccine within 30 days before enrollment.
12. The investigator considers that the patient has other reasons for not being suitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2022-09-24 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | from the first dose to within 30 days after the last dose.
  Adverse events evaluated by NCI CTCAE v5.0

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | within 42 days after the first dose
  One of Pharmacokinetic (PK) parameters.
Time to maximum concentration (Tmax) | within 42 days after the first dose
  One of Pharmacokinetic (PK) parameters.
Area under the curve (AUC) | within 42 days after the first dose
  One of Pharmacokinetic (PK) parameters.
Half-life (t1/2) | within 42 days after the first dose
  One of Pharmacokinetic (PK) parameters.
Clearance (CL) | within 42 days after the first dose
  One of Pharmacokinetic (PK) parameters.
Objective response rate | From the first dose to the date of disease progression or date of death from any cause, whichever comes first，up to 24months.
  the proportion of patients who have a Complete Response or Partial Response
Disease control rate | From the first dose to the date of disease progression or date of death from any cause, whichever comes first，up to 24months.
  the proportion of patients who have a Complete Response, Partial Response or Stable disease.

CONTACTS AND LOCATIONS:
Overall Officials: Hanying Bao, PhD, Study Director — Shanghai YingLi Pharmaceutical Co. Ltd.
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China